CLINICAL TRIAL: NCT06284629
Title: PD-DigiCare: Enhancing Referral Decision-making for Advanced Treatment in Parkinson's Disease Through Objective Measurements and Patient Reported Outcomes - a Multicentre Randomized Controlled Trial.
Brief Title: Enhancing Referral Decision-making for Advanced Treatment in Parkinson's Disease Through Objective Measurements and Patient Reported Outcomes.
Acronym: PD-DigiCare
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Bo Biering-Soerensen, MD, MPG, associate professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PD-DigiCare
Record Dates: First submitted 2024-02-14; First posted 2024-02-29 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: Wearable Devices; Objective measurements; Advanced treatment; Digital health
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Masking Description: Participants and physicians will be blinded to device and app data in the control group. Blinding of the group allocation is not possible due to the investigated device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of a wrist-worn wearable sensor that tracks motor symptoms and an app for patient-reported outcomes.
  Interventions: Device: Neptune
- Standard of Care (Active Comparator): The control group will wear the wrist-worn wearable sensor, but not be able to view the tracked data. They will report symptoms in the app, but the patient-reported outcomes won't be included in the clinical visits during the trial
  Interventions: Other: Standard clinical care

INTERVENTIONS:
Device: Neptune — Neptune is a software algorithm that utilizes data from wrist-worn sensors to track Parkinson motor symptoms and displays them in an easy to understand graph. Neptune Care is a mobile app that includes a patient portal, where patients can self-report symptoms, view their motor data and get medication reminders, and a physician portal, where the treating physician can view the objective motor data and patient-reported outcomes prior to a clinical visit.
  Other Names: Neptune Care
  Arms: Intervention
Other: Standard clinical care — Treatment and management according to standard clinical care
  Arms: Standard of Care

SUMMARY:
The overall aim of the trial is to compare the efficacy of using wearables and patient-reported outcome measures versus standard care in enhancing the timeliness of referrals to advanced monitoring of treatments for people with Parkinson's Disease.

DETAILED DESCRIPTION:
The study is a multicentre, parallel group, randomized controlled trial, investigating the value of using wearable devices and electronic patient-reported outcome measurements to improve clinical decision-making related to people with Parkinson's Disease.

Data from a wearable device and a mobile app will be compared to current standard of care.

90 participants will be recruited from the uptake area of the Movement Disorder Clinics (MDC) at Rigshospitalet Glostrup (RHG) and Odense University Hospital (OUH), as well as from 5 private practice neurologists in Denmark. They will equally be randomized to one of two groups: Intervention or Standard of Care.

Each participant will take part of the trial for one year, in which they will have 5 study visits:

* Baseline
* Clinical visits every 3 months (months 3, 6 and 9)
* Final visit after 12 months

They will be asked to wear the device and report symptoms in the app for one year. We will then compare decisions made related to changes in medication and referrals to advanced treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Idiopathic Parkinson's Disease
* Taking five or more doses of levodopa daily
* Experiencing fluctuations in motor function with regards to OFF time and/or dyskinesia.
* Able to utilize a digital product, either alone or assisted by a caregiver.

Exclusion Criteria:

* Consistent use of a wheelchair or walker which may interfere significantly with the remote monitoring of PD motor symptoms.
* Lack of understanding and proficiency in the Danish language.
* Inability to use wearable devices due to non-compliance, physical and/or skin sensitivity.
* Suffering from severe psychiatric disorders.
* Otherwise not qualified to receive advanced treatment (e.g., advanced cancer, severe heart failure).
* Already undergoing advanced treatment.
* Diagnosed with atypical or secondary parkinsonism.
* Other patient groups otherwise deemed ineligible by the project manager.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Differences between groups in algorithm-based motor symptom burden (time spent in the ON state without dyskinesias) at referral to evaluation for advanced treatment. | 1 year
  Time spent in the ON state without dyskinesias, as measured by the Neptune algorithm

SECONDARY OUTCOMES:
Differences in questionnaire data from baseline (inclusion visit) to end-of-intervention. | 1 year
  Global Sleep Assessment Scale (GSAQ). Every question is scored from 0-3 (highest worst)
Differences in questionnaire data from baseline (inclusion visit) to end-of-intervention. | 1 year
  Non-Motor Symptom Scale (NMSS). Scored from 0-360 (highest worst)
Changes in type of, frequency and dose of medication (calculated Levodopa Equivalent Dose, LED, by use of Tomlinson's scale) | 1 year
  Levodopa Equivalent Dose, LED, by use of Tomlinson's scale.
Differences in questionnaire data from baseline (inclusion visit) to end-of-intervention. | 1 year
  Movement Disorders Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Scored from 0-52 (UPDRS-II), 0-132 (UPDRS-III) and 0-44 (UPDRS-IV) (highest worst)
Differences in questionnaire data from baseline (inclusion visit) to end-of-intervention. | 1 year
  Parkinson's Disease Questionnaire (PDQ-39). Scored from 0-100 (highest worst)
Differences in questionnaire data from baseline (inclusion visit) to end-of-intervention. | 1 year
  EuroQol Questionnaire (EQ5D-5L). Scored from 0-1 and 0-100 (highest best).
Differences in questionnaire data from baseline (inclusion visit) to end-of-intervention. | 1 year
  Patient Global Impressions Scale - Improvement score (measurements of QoL) (PGI-I). Every question is scored from 1-7 (highest worst)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Biering-Soerensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Study data will be published in anonymized format as supplementary material to publications. Study protocol, SAP, ICF and analytic code will be available upon request.
Supporting Information: Study Protocol
Time Frame: Data will be published as supplementary material to publications.